CLINICAL TRIAL: NCT04606043
Title: Evaluation of the Effectiveness of Enamel Surface Treatment Using Sandblasting on the Bond Strength in the Rebonding Process: a Randomized Controlled Trial
Brief Title: Evaluation of the Sandblasting on the Rebonding Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UADS-2020-01
Record Dates: First submitted 2020-10-25; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Orthodontic Appliance Complication
MeSH Terms: interventions — Acid Etching, Dental

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sandblasting (Experimental): The enamel surfaces will be subjected to sandblasting prior to acid etching
  Interventions: Procedure: Sandblasting
- Acid Etching Alone (Active Comparator): Acid etching will be applied alone before the rebounding procedures
  Interventions: Procedure: Acid Etching

INTERVENTIONS:
Procedure: Sandblasting — Sandblasting will be applied onto the vestibular surfaces of the teeth before applying the etchant.
  Arms: Sandblasting
Procedure: Acid Etching — Only acid etching will be applied onto the vestibular surfaces of the teeth before rebonding
  Arms: Acid Etching Alone

SUMMARY:
Patients at the Orthodontic Department of University of Aleppo Dental School will be selected if they meet the inclusion criteria then fixed orthodontic treatment with 0.018-inch slot MBT appliances will be applied for those patients.

The aim of this study is to compare Two rebonding procedures by applying a split-mouth design. The clinical failure rates of the two rebonding procedures will be evaluated.

DETAILED DESCRIPTION:
The sample of this study will be chosen after examination of patients referred to the Department of Orthodontics at the University of Aleppo Dental School then subjects who meet the inclusion criteria will be included in this trial.

An information sheet will be given to each possible candidate. Then consent forms will be obtained.

All patients will receive both rebonding procedures by applying split-mouth design. Each patient will be asked to select an opaque sealed envelope from a box with 20 ones. Ten envelopes will Include instructions for applying sandblasting prior to acid-etching on the right upper premolars and acid-etching alone on the left upper premolars. In contrast, the other ten envelopes will include opposite instructions.

A total sample of 80 premolars will be obtained to study the clinical failure rates of the two rebonding procedures.

The 80 premolars will be randomly divided into two groups:

* The first group in which the enamel will be prepared using sandblasting prior to acid-etching.
* The second group in which the enamel will be prepared using acid-etching alone.

ELIGIBILITY:
Inclusion Criteria:

1. good general health and oral hygiene
2. willing and able to comply with the trial procedures
3. No crossbite, scissor bite, or occlusal interferences with the bonded/rebonded brackets in the premolars region (to prevent any potential early bond failure)
4. no craniofacial anomalies.

Exclusion Criteria:

1. any type of pervious orthodontic therapy
2. any need for ortho-surgical treatment or teeth extraction.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06-20 (Actual); Primary Completion 2012-05-10 (Actual); Study Completion 2012-06-15 (Actual)

PRIMARY OUTCOMES:
Bonding Failure Rate | After six month exactly of bonding the brackets onto the surfaces of the teeth
  Number of brackets loosing their bond to the enamel during the observation period divided by the total number of braces being applied.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Rami Dirie, DDS MSc, Principal Investigator — Specialist and Clinical Lecturer, Department of Orthodontics, University of Aleppo; Heba M. Al-Ibrahim, DDS, Principal Investigator — MSc student in Orthodontics, University of Damascus; Jamal Dabbas, DDS MSc PhD, Study Director — Professor of Orthodontics, Department of Orthodontics, University of Aleppo; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Professor of Orthodontics, Department of Orthodontics, University of Damascus
Locations (1):
- Department of Orthodontics, University of Aleppo Dental School, Aleppo, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egan FR, Alexander SA, Cartwright GE. Bond strength of rebonded orthodontic brackets. Am J Orthod Dentofacial Orthop. 1996 Jan;109(1):64-70. doi: 10.1016/s0889-5406(96)70164-6. PMID 8540484
- [Background] Bishara SE, Laffoon JF, Vonwald L, Warren JJ. The effect of repeated bonding on the shear bond strength of different orthodontic adhesives. Am J Orthod Dentofacial Orthop. 2002 May;121(5):521-5. doi: 10.1067/mod.2002.123042. PMID 12045771
- [Background] Faust JB, Grego GN, Fan PL, Powers JM. Penetration coefficient, tensile strength, and bond strength of thirteen direct bonding orthodontic cements. Am J Orthod. 1978 May;73(5):512-25. doi: 10.1016/0002-9416(78)90241-5. No abstract available. PMID 354405
- [Background] Mizrahi E. Success and failure of banding and bonding. A clinical study. Angle Orthod. 1982 Apr;52(2):113-7. doi: 10.1043/0003-3219(1982)0522.0.CO;2. PMID 7049010
- [Derived] Dirie AR, Hajeer MY, Dabbas J, Al-Ibrahim HM. Evaluation of sandblasting with acid etching versus acid etching alone in the preparation of enamel for rebonding orthodontic brackets: An in vitro study and a randomized controlled trial. J World Fed Orthod. 2021 Mar;10(1):3-8. doi: 10.1016/j.ejwf.2020.12.001. Epub 2021 Jan 7. PMID 33422476